CLINICAL TRIAL: NCT04268225
Title: Ultrasound Guided Peripheral Intravenous Catheterization in Children Hospitalized in the Pediatric Intensive Care Unit: a Randomized Controlled Prospective Trial.
Brief Title: Ultrasound Guided Peripheral Intravenous Catheterization in the Pediatric Intensive Care Unit.
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Rabin Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 0044-20-RMC
Record Dates: First submitted 2020-02-09; First posted 2020-02-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-02

CONDITIONS: Peripheral Venous Cannulation

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ultrasound Guided Dynamic Needle Tip Positioning Technique (Experimental): In this arm the US transducer, protected with a sterile cover and sterile gel will be placed in the short axis above the distal end of the selected vein, moving the probe to place the vein in the center of the ultrasound screen under the middle mark of the image. The catheter needle will be inserted close to the transducer. The needle tip will be visualized as a white dot on the ultrasound screen. Then, the transducer will be shifted slightly proximally until the white dot disappears from the screen. The needle and the transducer will be moved alternately toward the patient several times to visualize the needle tip in real time. After penetrating the anterior wall of the vein, these steps will be repeated a few more times with a smaller insertion angle to visualize the white dot in the vein. Finally, the outer catheter will be fully advanced and the needle core will be extracted.
  Interventions: Procedure: US guided dynamic needle tip positioning peripheral intravenous cannulation
- Traditional insertion group (Active Comparator): For traditional insertion technique insertion attempt will be blind or tactile. Otherwise, the same protocol and measurements as elaborated for the US guided group will be applied.
  Interventions: Procedure: Traditional peripheral intravenous cannulation

INTERVENTIONS:
Procedure: US guided dynamic needle tip positioning peripheral intravenous cannulation — Catheterizations will be performed by one of three pediatric intensivists with vast experience in both traditional and US guided DNTP techniques for peripheral intravenous access. The operator will be allowed to independently choose which peripheral vein to cannulate. If necessary, patients will be given supplemental dose of sedation and analgesia in addition to the already given continuous infusions for invasive mechanical ventilation. Before puncture, the limb will be taped and maintained in an optimal position. A tourniquet will be placed proximal to the planned cannulation site. The site of puncture will be disinfected with Chlorhexidine gluconate 0.5% w/v, Alcohol 70% v/v. The choice of catheter will be left to the discretion of the operator. Available PIV cannulas include : 14 GA, 2X45 mm; 17 GA, 1.4X45 mm; 18 GA 1.2X45 mm; 20 GA 1X32mm BD Venflon™ and 24 GA, 0.7X19 mm; 26 GA 0.6X19 mm BD Neoflon™ (Becton Dickinson Infusion Therapy AB, Helsingborg, Sweden).
  Arms: Ultrasound Guided Dynamic Needle Tip Positioning Technique
Procedure: Traditional peripheral intravenous cannulation — For traditional insertion technique insertion attempt will be blind or tactile.
  Arms: Traditional insertion group

SUMMARY:
This is a randomized controlled prospective study. The purpose of this study is to compare a recently described technique of ultrasound (US) guided, dynamic needle tip positioning (DNTP), to the traditional technique of vein visualization and palpation for peripheral venous cannulation in intubated, sedated, and mechanically ventilated pediatric intensive care unit (PICU) patients. First attempt success rate, overall success rate within 3 attempts or 10 minutes (whichever comes first), number of attempts to success, time to success and cannula sizes will be compared between the 2 techniques. The study will include intubated, sedated and mechanically ventilated children, aged 0-18 years, hospitalized in the PICU who require peripheral intravenous (PIV) access for their management.

ELIGIBILITY:
Inclusion Criteria:

1. Invasively ventilated
2. Younger than 18 years
3. Peripheral venous access required
4. Difficult intravenous access (DIVA) score of 4 or greater (on a scale of 0-10 with higher scores implying more difficult access)

Exclusion Criteria:

1. Refusal to consent
2. Research staff not available

Max Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 90 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2022-03 (Estimated); Study Completion 2022-03 (Estimated)

PRIMARY OUTCOMES:
Success of peripheral IV cannulation on first attempt | 10 minutes
  Assessment of peripheral IV cannulation success on first attempt (Yes vs No)

SECONDARY OUTCOMES:
Overall peripheral IV cannulation success rate | 10 minutes
  The overall success rate of peripheral intravenous cannulation within 3 attempts.
Time to successful peripheral IV cannulation | up to 10 minutes
  Defined as the time from first skin puncture to successful cannulation (minutes).
Number of attempts to success | up to 10 minutes
  Number of puncture attempts (1,2 or 3) needed for achieving a a successful cannulation
Inserted cannula diameter | up to 10 minutes
  Cannula diameter (in GA) successfully inserted

OTHER OUTCOMES:
Patient age | 1 day (At the time of peripheral IV cannulation)
  Age in years
Patient sex | 1 day (At the time of peripheral IV cannulation)
  Female vs Male
Patient body mass index (BMI) | 1 day (At the time of peripheral IV cannulation)
  BMI (in kg/m^2) for age percentile
Patient inotropic and vasoactive support | 1 day (At the time of peripheral IV cannulation)
  Vasoactive-Inotropic Score (VIS score)
Admission-cannulation time | 1 day (At the time of peripheral IV cannulation)
  Time from hospital admission to first attempt of cannulation
Reason for admission | 1 day (At the time of peripheral IV cannulation)
  Medical vs Surgical

CONTACTS AND LOCATIONS:
Overall Officials: Avichai Weissbach, MD, Principal Investigator — Rabin Medical Center

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Costantino TG, Parikh AK, Satz WA, Fojtik JP. Ultrasonography-guided peripheral intravenous access versus traditional approaches in patients with difficult intravenous access. Ann Emerg Med. 2005 Nov;46(5):456-61. doi: 10.1016/j.annemergmed.2004.12.026. PMID 16271677
- [Background] Doniger SJ, Ishimine P, Fox JC, Kanegaye JT. Randomized controlled trial of ultrasound-guided peripheral intravenous catheter placement versus traditional techniques in difficult-access pediatric patients. Pediatr Emerg Care. 2009 Mar;25(3):154-9. doi: 10.1097/PEC.0b013e31819a8946. PMID 19262420
- [Background] Otani T, Morikawa Y, Hayakawa I, Atsumi Y, Tomari K, Tomobe Y, Uda K, Funakoshi Y, Sakaguchi C, Nishimoto S, Hataya H. Ultrasound-guided peripheral intravenous access placement for children in the emergency department. Eur J Pediatr. 2018 Oct;177(10):1443-1449. doi: 10.1007/s00431-018-3201-3. Epub 2018 Jun 30. PMID 29961178
- [Background] Vinograd AM, Zorc JJ, Dean AJ, Abbadessa MKF, Chen AE. First-Attempt Success, Longevity, and Complication Rates of Ultrasound-Guided Peripheral Intravenous Catheters in Children. Pediatr Emerg Care. 2018 Jun;34(6):376-380. doi: 10.1097/PEC.0000000000001063. PMID 28221281
- [Background] Elkhunovich M, Barreras J, Bock Pinero V, Ziv N, Vaiyani A, Mailhot T. The use of ultrasound for peripheral IV placement by vascular access team nurses at a tertiary children's hospital. J Vasc Access. 2017 Jan 18;18(1):57-63. doi: 10.5301/jva.5000615. Epub 2016 Nov 15. PMID 27886365
- [Background] Benkhadra M, Collignon M, Fournel I, Oeuvrard C, Rollin P, Perrin M, Volot F, Girard C. Ultrasound guidance allows faster peripheral IV cannulation in children under 3 years of age with difficult venous access: a prospective randomized study. Paediatr Anaesth. 2012 May;22(5):449-54. doi: 10.1111/j.1460-9592.2012.03830.x. Epub 2012 Mar 12. PMID 22409596
- [Background] Kiberenge RK, Ueda K, Rosauer B. Ultrasound-Guided Dynamic Needle Tip Positioning Technique Versus Palpation Technique for Radial Arterial Cannulation in Adult Surgical Patients: A Randomized Controlled Trial. Anesth Analg. 2018 Jan;126(1):120-126. doi: 10.1213/ANE.0000000000002261. PMID 29135593
- [Background] Liu L, Tan Y, Li S, Tian J. "Modified Dynamic Needle Tip Positioning" Short-Axis, Out-of-Plane, Ultrasound-Guided Radial Artery Cannulation in Neonates: A Randomized Controlled Trial. Anesth Analg. 2019 Jul;129(1):178-183. doi: 10.1213/ANE.0000000000003445. PMID 29787409
- [Background] Takeshita J, Inata Y, Ito Y, Nishiyama K, Shimizu Y, Takeuchi M, Shime N. Dynamic Needle Tip Positioning for Ultrasound-Guided Placement of a Peripherally Inserted Central Catheter in Pediatric Patients. J Cardiothorac Vasc Anesth. 2020 Jan;34(1):114-118. doi: 10.1053/j.jvca.2019.04.029. Epub 2019 May 2. PMID 31129072
- [Background] Takeshita J, Yoshida T, Nakajima Y, Nakayama Y, Nishiyama K, Ito Y, Shimizu Y, Takeuchi M, Shime N. Dynamic Needle Tip Positioning for Ultrasound-Guided Arterial Catheterization in Infants and Small Children With Deep Arteries: A Randomized Controlled Trial. J Cardiothorac Vasc Anesth. 2019 Jul;33(7):1919-1925. doi: 10.1053/j.jvca.2018.12.002. Epub 2018 Dec 4. PMID 30638922
- [Background] Takeshita J, Yoshida T, Nakajima Y, Nakayama Y, Nishiyama K, Ito Y, Shimizu Y, Takeuchi M, Shime N. Superiority of Dynamic Needle Tip Positioning for Ultrasound-Guided Peripheral Venous Catheterization in Patients Younger Than 2 Years Old: A Randomized Controlled Trial. Pediatr Crit Care Med. 2019 Sep;20(9):e410-e414. doi: 10.1097/PCC.0000000000002034. PMID 31232853